CLINICAL TRIAL: NCT04912336
Title: Extra Corporeal Life Support and Modification of Hemostasis
Brief Title: Extracorporeal Life Support and Modification of Hemostasis
Acronym: ELMOH
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-07099
Record Dates: First submitted 2021-05-06; First posted 2021-06-03 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Bleeding Disorder; Extra Corporeal Life Support; Thrombosis
MeSH Terms: conditions — Hemostatic Disorders; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood tests for coagulation parameters
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VV-ECMO: Patients supported because of respiratory failure by Veno-Venous Extra Corporeal Membrane Oxygenator.
  Interventions: Diagnostic Test: Standard coagulation profile; Diagnostic Test: Specific coagulation tests; Other: Bleeding Scores
- VA-ECMO: Patients supported because of circulatory failure by Veno-Arterial Extra Corporeal Membrane Oxygenator.
  Interventions: Diagnostic Test: Standard coagulation profile; Diagnostic Test: Specific coagulation tests; Other: Bleeding Scores

INTERVENTIONS:
Diagnostic Test: Standard coagulation profile — prothrombin time (PT), international normalized ratio (INR), activated partial thromboplastin time (aPTT), the fibrinogen level, plateletcount
Diagnostic Test: Specific coagulation tests — AT III, anti Xa, ACT, ROTEM
Other: Bleeding Scores — Global Utilization of Streptokinase and Tpa for Occluded arteries definition of bleeding (GUSTO) AND Bleeding Academic Research Consortium Definition for Bleeding (BARC)

SUMMARY:
To evaluate change in coagulation tests during a 48-h period after initiation VV-ECMO and VA-ECMO.

(ECMO= Extra Corporeal Membrane Oxygenator) Assessment of bleeding during Veno-Venous Extracoporeal Membrane Oxygenator (VV-ECMO) and Veno-Arterial Extracoporeal Membrane Oxygenator (VA-ECMO).

DETAILED DESCRIPTION:
This is a multi-center, prospective, pilot cohort study, performed in the Intensive Care Units (ICUs) of the Ghent University Hospital, CHU Liège, University Hospital Brussels, and University Hospital Munster.

Each group will contain 20 subjects; in total there will be 40 subjects 2 groups of 20 patients GROUP 1: VV-ECMO n = 20 GROUP 2: VA-ECMO n = 20

* Demographics: age, sex, comorbidities, medication, reason for ECMO therapy
* Simplified Acute Physiology Score (SAPS) 3 at time of ICU admission.
* Components of the Sequential Organ Failure Assessment score daily (based on worst value of each component of the score)
* ECMO characteristics (place of cannulation, type of cannulas, oxygenator, bloodflow, gasflow and pressure registrations)
* Incidence and severity of bleeding, scored according to the GUSTO and BARC scores
* Coagulation profile: At inclusion (before heparine infusion is started), 2h after start of therapy, 24h, and 48h, and at specific moments of clinical suspicion of profound altered hemostasis. We defined a coagulation profile as a set of tests that includes

  * prothrombin time (PT), international normalized ratio (INR)
  * activated partial thromboplastin time (aPTT) and heparin ratio
  * the fibrinogen level
  * platelets
  * ACT (iACT®, …)
  * D-dimer
  * ROTEM (extem, intem, heptem) or TEG (Utrecht)
  * AT III
  * anti Xa
* Temperature daily (H/L) (core)
* Patient characteristics that may influence coagulation or the results of coagulation tests: body weight, Body Mass Index, drugs, C-reactive protein (as a marker for inflammation), Hemoglobin level, LDH, unconjugated bilirubin, (or haptoglobine or plasma free haemoglobin, if tested)
* Heparin dose

ELIGIBILITY:
Inclusion Criteria:

* GROUP 1: patients who will be initiated on VV-ECMO within a 12-h period
* GROUP 2: patients who will be initiated on VA-ECMO within a 12-h period
* ≥ 18 years
* Signed Informed Consent, signed by subject or authorized representative

Exclusion criteria:

Expected survival <48-h Known coagulopathy Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * GROUP 1: patients who will be initiated on VV-ECMO within a 12-h period
  * GROUP 2: patients who will be initiated on VA-ECMO within a 12-h period
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Thrombocytopenia | 48 hours
  Moderate thrombocytopenia lower than 150 x 103/µL in 25% of recruited patients

SECONDARY OUTCOMES:
Bleeding problems, Type 2 Bleeding according to BARC criteria or moderate bleeding according to GUSTO criteria | 48 hours
  incidence of clinical overt bleeding
Clotting problems | 48 hours
  Incidence of deep venous trombosis or emboli or ECMO circuit problems due to clotting
Need for transfusion | 48 hours
  Need for transfusion of packed red blood cells
Change in visco-elastic testing | At 2 hours, 24 hours, 48 hours
  ROTEM changes
Survival | 1 year
  survival in the ICU, in the hospital, at day 28, day 90, 6months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Harlinde Peperstraete, MD, Principal Investigator — University Hospital, Ghent
Locations (6):
- Belgium (5):
  - CHU Charleroi, Lodelinsart, Henegouwen
  - CHU UCL Namur- Godinne, Yvoir, Namen
  - Ghent University Hospital, Ghent
  - University Hospital Brussels, Jette
  - Centre Hospitalier Universitaire Liege, Liège
- University Hospital Münster, Münster, Germany

IPD SHARING:
Plan to Share IPD: Undecided
All data will be put in Redcap. At inclusion, at inclusion +2h, at inclusion +24 and at inclusion +48h: a clotting panel and clinical observation about bleedina and clotting will be performed.